CLINICAL TRIAL: NCT01468272
Title: A Single-dose,Open-label,Randomized,2-way Cross-over,Clinical Pharmacology Study of CHF1535 50/6 NEXT DPI® Fixed Combination of Beclomethasone Dipropionate 50µg Plus Formoterol Fumarate 6µg)Versus the Free Combination of Licensed Beclomethasone DPI and Formoterol DPI in Asthmatic Children
Brief Title: Clinical Pharmacology of CHF 1535 50/6 ug Next DPI in Children 5-11 Years Old
Acronym: PAED4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-1103-PR-0058
Record Dates: First submitted 2011-10-28; First posted 2011-11-09 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Asthma in Children
Keywords: asthma children NEXT DPI LABA ICS inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- reference treatment (Active Comparator): Free combination of Beclomethasone dipropionate DPI and Formoterol fumarate DPI
  Interventions: Drug: free comb. beclomethasone DPI and formoterol DPI
- CHF 1535 NEXT DPI (Experimental): CHF 1535 50/6 NEXT DPI
  Interventions: Drug: CHF 1535 50/6 NEXT DPI

INTERVENTIONS:
Drug: free comb. beclomethasone DPI and formoterol DPI — free combination of beclomethasone dipropionate 100 ug/unit DPI (two inhalations, total dose 200 ug), and formoterol fumarate 6 ug/unit DPI (four inhalations, total dose 24 ug).
  Arms: reference treatment
Drug: CHF 1535 50/6 NEXT DPI — four inhalations of CHF 1535 50/6 NEXT DPI, a fixed combination of beclomethasone dipropionate 50 ug plus formoterol fumarate 6 ug (TOTAL DOSE:BDP/FF 200/24 ug)
  Arms: CHF 1535 NEXT DPI

SUMMARY:
This is a pharmacokinetic comparison of CHF 1535 50/6 NEXT DPI versus the free combination of Beclomethasone DPI and Formoterol DPI in children (5 to 11 years old) of a formulation already approved in adults.

DETAILED DESCRIPTION:
Pharmacokinetic study in asthmatic children 5 to 11 years old treated with either a fixed combination of beclomethasone 50 ug/unit dose plus formoterol fumarate 6 ug/unit dose via the NEXT DPI dry powder inhaler or a free combination of Beclomethasone 100 ug DPI and Formoterol 6 ug DPI according to a cross-over design.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female children aged 5 -11y
2. Written informed consent obtained by parents/legal representative (according to local regulation) and by the minor (age and local regulation permitting).
3. Children with stable asthma
4. Children with asthma on regular treatment with ICS or using short-acting inhaled beta2-agonists as reliever to control asthma symptoms
5. Forced expiratory volume in one second (FEV1) > 70% of predicted values (% pred) after withholding beta2-agonists treatment for a minimum of 4 h prior to each study treatment.
6. A cooperative attitude and ability to be trained about the proper use of DPI and compliant to study procedures.

Exclusion Criteria:

1. Past or present diagnoses of cardiovascular, renal or liver disease
2. Known hypersensitivity to the active treatments
3. Exacerbation of asthma symptoms within the previous 4 weeks
4. Inability to perform the required breathing technique and blood sampling
5. Hospitalization due to exacerbation of asthma within 1 month prior to screening (visit 1)
6. Lower respiratory tract infection within 1 month prior to screening (visit 1)
7. Disease (other than asthma) which might influence the outcome of the study
8. Obesity, i.e. > 97% weight percentile by local standards

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
B17MP (active metabolite of BDP) Area Under Curve (AUC) | predose, 15,30min, 1,2,4,6,8 hours post dose
  B17MP: Profile of Pharmacokinetics

SECONDARY OUTCOMES:
B17MP Cmax,Tmax,T1/2 | predose, 15min,30min,1,2,4,6,8 hours post dose
  BDP: profile of pharmacokinetics.
BDP Area Under Curve (AUC), Cmax, Tmax, T1/2 | predose, 15min,30min,1,2,4,6,8 hours postdose
  BDP: profile of Pharmacokinetics
Formoterol Area Under Curve (AUC), Cmax, Tmax, T1/2 | predose, 15min, 30 min, 1,2,4,6,8 hours postdose
  Formoterol: profile of pharmacokinetics
plasma potassium Area Under Curve (AUC), Cmin, Tmin | predose, 15min, 30min, 1, 2, 4, 6, 8 hours postdose
  plasma potassium to evaluate drug systemic effect
Heart Rate: Time averaged Heart Rate value: AUC0-t/t | predose, 15min, 30min, 1, 2, 4, 6, 8 hours postdose
  Heart Rate to evaluate drug systemic effect
Urinary Cortisol: Amount excreted in 0-8hours (Ae),8h cortisol urinary excretion normalized for 8h creatinine excretion (Ae/Aecreat). | from predose up to 8 hours postdose
  Urinary cortisol to evaluate drug systemic effect

CONTACTS AND LOCATIONS:
Overall Officials: Hans Bisgaard, Principal Investigator — BorneAstmaKlinikken, Copenaghen, Denmark
Locations (1):
- BørneAstmaKlinikken, Hans Knudsens Plads 1A,, Copenhagen, Denmark

REFERENCES:
- [Result] Chawes BL, Govoni M, Kreiner-Moller E, Vissing NH, Poorisrisak P, Mortensen L, Nilsson E, Bisgaard A, Dossing A, Deleuran M, Skytt NL, Samandari N, Piccinno A, Sergio F, Ciurlia G, Poli G, Acerbi D, Singh D, Bisgaard H. Systemic exposure to inhaled beclometasone/formoterol DPI is age and body size dependent. Respir Med. 2014 Aug;108(8):1108-16. doi: 10.1016/j.rmed.2014.05.007. Epub 2014 Jun 17. PMID 24993817
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2011-001208-36